CLINICAL TRIAL: NCT01430182
Title: Intraoperative Methadone Versus Morphine for Postoperative Pain Control in Patients Undergoing Intramedullary Nailing or Open Reduction and Internal Fixation of the Tibia
Brief Title: Intraoperative Methadone vs Morphine for Postoperative Pain Control in Patients Undergoing Surgery of the Tibia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Shortages of study drug, difficulty enrolling patients
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Neil S Bailard, Assistant Professor, Department of Anesthesiology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-28734
Record Dates: First submitted 2011-09-06; First posted 2011-09-08 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Pain, Postoperative
Keywords: Adult; Female; Humans; Intraoperative Care/methods; Male; Methadone/administration & dosage; Analgesics/therapeutic use; Methadone/therapeutic use; Morphine/therapeutic use; Middle Aged; Pain Measurement/drug effects; Pain Measurement/methods; Pain, Postoperative/prevention & control; Prospective Studies; Double-Blind Method; Tibial Fractures/surgery; Young Adult; Orthopedics
MeSH Terms: conditions — Pain, Postoperative; Pain; Tibial Fractures | interventions — Methadone; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone 0.2 mg/kg (Experimental): 0.2 mg/kg methadone by actual body weight, administered over ten minutes, initiated after induction of anesthesia and endotracheal intubation complete.
  Interventions: Drug: Methadone
- Morphine 0.2 mg/kg (Active Comparator): 0.2 mg/kg morphine by actual body weight, administered over ten minutes, initiated after induction of anesthesia and endotracheal intubation complete.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Methadone — 0.2 mg*kg-1 by actual body weight, administered over 10 minutes, once induction of anesthesia and endotracheal intubation are complete.
  Other Names: Bioniche Pharma, METHADONE HYDROCHLORIDE INJECTION
  Arms: Methadone 0.2 mg/kg
Drug: Morphine — 0.2 mg*kg-1 by actual body weight, administered over 10 minutes, once induction of anesthesia and endotracheal intubation are complete.
  Other Names: Morphine sulfate
  Arms: Morphine 0.2 mg/kg

SUMMARY:
The purpose of this study is to determine whether, for surgery of the tibia, one dose of methadone provides better control of pain afterward as compared to morphine, which is the usual drug given to control pain after surgery. Immediately after the beginning of general anesthesia ("intraoperatively"), subjects will receive one dose of either methadone or morphine, in the amount of 0.2 milligrams per kilogram of body weight, intravenously.

The primary hypothesis is that, subjects who receive one dose of methadone intraoperatively will require less pain medicine than subjects who receive one dose of morphine intraoperatively.

DETAILED DESCRIPTION:
Satisfactory pain control can generally be achieved after major surgery of the tibia through a combination of enteral and parenteral medications, neuraxial techniques (such as epidural analgesia), and/or regional techniques (such as sciatic and femoral nerve block). Intramedullary nailing (IMN) and open reduction/internal fixation (ORIF) of the tibia have been important exceptions, and postoperative pain control can be difficult to achieve in these cases.

Surgical repair of fractures of the tibial shaft and of the proximal tibia can be complicated by compartment syndrome, with the possibility of substantial morbidity and loss of function if not detected and treated promptly. It is not always possible to determine preoperatively which tibial fractures are at high risk, and which are low risk for this complication.

The hallmark of compartment syndrome, and often the earliest sign, is pain out of proportion to the nature of the injury. This pain is poorly relieved by morphine or other strong analgesics. In contrast, because peripheral nerve blocks, spinals, and epidurals can completely block the neural transmission of nociceptive stimuli, they can obliterate this important early warning sign. For this reason, orthopedic surgeons often request of anesthesiologists that patients who are to undergo IMN or ORIF of at-risk tibial fractures not receive neuraxial blocks or regional nerve blocks. As a result, patients who undergo IMN/ORIF of the tibia often receive poor pain relief because they are denied these treatment options, even though the vast majority do not go on to develop compartment syndrome.

A typical postoperative pain regimen for IMN/ORIF tibia patients usually begins with a parenteral opioid such as morphine, along with an oral analgesic such as acetaminophen/hydrocodone ("Vicodin"), acetaminophen/codeine ("Tylenol #3"), or tramadol. The parenteral opioid is often given by patient-controlled analgesia pump (PCA), with supplemental doses ordered for breakthrough pain. A major disadvantage of morphine is its equilibration half-time of 2-4 hours. Thus there is considerable lag between the plasma morphine concentration (which peaks immediately) and the morphine concentration at the effector sites. This hysteresis results in the slow onset of analgesia, with peak analgesia occurring some 80-90 minutes after IV administration. It can also result in excessive somnolence, when several demand doses in a row finally take effect. Morphine has an elimination half-time of 2-3 hours. These repeated bolus doses result in the classic "see-saw" graph of plasma morphine concentration over time, with its peaks and troughs. Methadone, in contrast, has a much lower equilibration half-time, on the order of 4-8 minutes. This results in quicker transfer of methadone from the plasma to its effector sites, and hence quicker onset of action, with peak analgesia occurring in just 11.3 minutes. Methadone's elimination half-life after a single dose is approximately 24-36 hours, resulting in prolonged analgesia, with less re-dosing necessary.

Most recently, for multilevel thoracolumbar spine surgery with instrumentation and fusion, intraoperative intravenous methadone was shown to have substantial opioid-sparing effects compared to intraoperative sufentanil bolus with sufentanil infusion, and similar rates of side effects such as hypotension, respiratory depression, hypoxemia, arrhythmia, nausea, and vomiting.

For these reasons, administering an intraoperative loading dose of 0.2 mg/kg methadone IV should result in better analgesia for ORIF and IMN of the tibia, compared with an intraoperative loading dose of 0.2 mg/kg morphine IV. This dose of methadone has previously been shown to yield plasma concentrations above the Minimum Effective Concentration, without excessive respiratory depression. This dose has been shown to provide long-lasting analgesia after painful procedures, often to the point that subjects needed no supplemental analgesics at all, or only non-narcotic analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled for elective, non-emergent intramedullary nailing (IMN) or open reduction/internal fixation (ORIF) of the tibia at Ben Taub General Hospital
* Able to give consent (not cognitively impaired or intoxicated)
* Subjects must be 18-50 years of age
* American Society of Anesthesiologists (ASA) physical status I-III
* Scheduled for primary intramedullary nailing or open reduction/internal fixation of fractures of the tibial shaft or proximal tibia. This must be the first operation for this injured extremity.
* Associated fractures of the fibula will be allowed.
* Minor lacerations or other associated injuries like "road rash" or open wounds requiring skin graft are permitted

Exclusion Criteria:

* Subjects who have taken preoperative opioids for more than 7 days before surgery (i.e., tolerant)
* Regular use of opioids (whether recreational/illicit or prescribed) within the six months before injury
* Subjects who are recommended to receive a regional nerve block or a neuraxial technique (spinal or epidural) by the attending orthopedic surgeon
* Subjects who refuse general anesthesia
* Subjects deemed to be moderately or severely hypovolemic
* External fixator already in place on the injured extremity
* Presence of other moderate-to-severe or distracting injuries, such as orthopedic, cervical spine, neurological, intra-abdominal, or intra-thoracic injuries. Minor abrasions/lacerations such as "road rash" or open wounds are acceptable. Associated fibular injuries are acceptable. Small peripheral injuries such as a finger or toe requiring percutaneous pinning are acceptable. Small skin grafts (no more than 100 cm^2) are permitted
* Pregnancy or breastfeeding (verify urine pregnancy test)
* Associated or pre-existing head injury or Traumatic Brain Injury
* Difficulty or inability to understand the study or the protocol
* Severe obesity (BMI > 36.0 kg/m^2)
* Known respiratory or cardiovascular problems, such as obstructive sleep apnea, or oxygen saturation of less than 96% on room air
* Acute bronchial asthma
* Chronic renal failure (serum creatinine > 2.0 mg/dL)
* Liver failure (defined as history of cirrhosis or fulminant hepatic failure)
* History of myocardial infarction or heart failure
* History of prolonged QT syndrome (QTc 450ms or more for men and 460ms or more for women)
* Known contraindications to methadone including hypothyroidism, Addison's disease, prostatic hypertrophy, or urethral stricture
* History of allergic reaction to morphine, methadone, acetaminophen, or hydrocodone
* Taking medications known to induce or inhibit the cytochrome p450 enzyme systems, such as azole antifungals, macrolide antibiotics, and selective serotonin reuptake inhibitors
* Taking antiretroviral medications (any)
* Consumption of grapefruit or grapefruit juice within past 5 days

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2011-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil S Bailard, MD, Principal Investigator — Dept. of Anesthesiology, Baylor College of Medicine
Locations (1):
- Ben Taub General Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538
- [Background] Gourlay GK, Willis RJ, Lamberty J. A double-blind comparison of the efficacy of methadone and morphine in postoperative pain control. Anesthesiology. 1986 Mar;64(3):322-7. doi: 10.1097/00000542-198603000-00004. PMID 3954126
- [Background] Gourlay GK, Willis RJ, Wilson PR. Postoperative pain control with methadone: influence of supplementary methadone doses and blood concentration--response relationships. Anesthesiology. 1984 Jul;61(1):19-26. PMID 6742480
- [Background] Gourlay GK, Wilson PR, Glynn CJ. Pharmacodynamics and pharmacokinetics of methadone during the perioperative period. Anesthesiology. 1982 Dec;57(6):458-67. doi: 10.1097/00000542-198212000-00005. No abstract available. PMID 6128949
- [Background] Gourlay GK, Wilson PR, Glynn CJ. Methadone produces prolonged postoperative analgesia. Br Med J (Clin Res Ed). 1982 Feb 27;284(6316):630-1. doi: 10.1136/bmj.284.6316.630. No abstract available. PMID 6802264

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were inpatients in Ben Taub General Hospital, a General and Teaching Hospital in Houston, Texas. Subjects were enrolled from October 2011 through May 2013.
Pre-assignment Details: 18 subjects were approached for participation. 1 was a screen failure, yielding 17 subjects who were randomized and received methadone or morphine
Period: Overall Study
Arm/Group | Methadone 0.2 mg/kg | Morphine 0.2 mg/kg
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methadone 0.2 mg/kg | Morphine 0.2 mg/kg | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (7.4) | 29.3 (10.2) | 30.7 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption
Description: Number of morphine equivalents used by subject during first 24 hours after discharge from Post-Anesthesia Care Unit
Time Frame: First 24 hours after discharge from Post-Anesthesia Care Unit
Measure: Mean (Standard Deviation); unit: mg of morphine IV equivalents
Arm/Group | Methadone 0.2 mg/kg | Morphine 0.2 mg/kg
Number analyzed (Participants) | 9 | 8
mg of morphine IV equivalents | 50.9 (38.7) | 37.5 (15.4)
Statistical Analysis 1: Comparison: Methadone 0.2 mg/kg vs Morphine 0.2 mg/kg; Test type: Superiority or Other; p = 0.37, t-test, 1 sided; unpaired

ADVERSE EVENTS:
Arm/Group | Methadone 0.2 mg/kg | Morphine 0.2 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 1/9 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methadone 0.2 mg/kg (N=9) | Morphine 0.2 mg/kg (N=8)
Excessive sedation or excessive somnolence (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Shortages of IV methadone prompted closure of trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No